CLINICAL TRIAL: NCT05323461
Title: A Randomized, Double-blind, and Positive-controlled Phase III Clinical Trial to Evaluate the Immunogenicity and Safety of SCTV01C (A Bivalent SARS-CoV-2 Trimeric Spike Protein Vaccine) and SCTV01E (A COVID-19 Alpha/Beta/Delta/Omicron Variants S-Trimer Vaccine) in Population Aged ≥18 Years Previously Vaccinated With Either Inactivated or mRNA COVID-19 Vaccine or Previously Diagnosed With COVID-19
Brief Title: A Study to Evaluate the Immunogenicity and Safety of Two Recombinant Protein COVID-19 Vaccines in Population Aged ≥18 Years as Booster Vaccines
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SCTV01C-E-01-UAE-1
Record Dates: First submitted 2022-04-10; First posted 2022-04-12 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: COVID-19; SARS-CoV-2; Vaccine
MeSH Terms: conditions — COVID-19 | interventions — SCTV01C vaccine; BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1: SCTV01C (Experimental): one dose of SCTV01C on D0
  Interventions: Biological: SCTV01C
- Cohort 1: SCTV01E (Experimental): one dose of SCTV01E on D0
  Interventions: Biological: SCTV01E
- Cohort 1: Active comparator (Active Comparator): one dose of Sinopharm inactivated COVID-19 vaccine on D0
  Interventions: Biological: Sinopharm inactivated COVID-19 vaccine
- Cohort 2: SCTV01C (Experimental): one dose of SCTV01C on D0
  Interventions: Biological: SCTV01C
- Cohort 2: SCTV01E (Experimental): one dose of SCTV01E on D0
  Interventions: Biological: SCTV01E
- Cohort 2: Active comparator (Active Comparator): one dose of Comirnaty on D0
  Interventions: Biological: Comirnaty

INTERVENTIONS:
Biological: SCTV01C — intramuscular injection
  Arms: Cohort 1: SCTV01C; Cohort 2: SCTV01C
Biological: SCTV01E — intramuscular injection
  Arms: Cohort 1: SCTV01E; Cohort 2: SCTV01E
Biological: Sinopharm inactivated COVID-19 vaccine — intramuscular injection
  Arms: Cohort 1: Active comparator
Biological: Comirnaty — intramuscular injection
  Arms: Cohort 2: Active comparator

SUMMARY:
The study is a randomized, double-blind, and positive-controlled Phase III booster study. It will evaluate the immunogenicity and safety of one dose of SCTV01C or SCTV01E as booster compared with either one dose of Sinopharm inactivated COVID-19 vaccine (Cohort 1) or one dose of Comirnaty (Cohort 2).

DETAILED DESCRIPTION:
Approximately 1,800 participants aged 18 years old and above will be enrolled in this study. 1,350 participants who previously received Sinopharm inactivated COVID-19 vaccine will be enrolled to Cohort 1. 450 participants who previously received mRNA COVID-19 vaccine or previously diagnosed with COVID-19 will be enrolled to Cohort 2.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years old when signing ICF;
2. For Subgroup 1 in Cohort 1: Participants who were previously vaccinated with 2 or 3 doses of Sinopharm inactivated COVID-19 vaccine. The interval between the date of last dose and the date of this study vaccination should be 3 to 24 months.

   For Subgroup 2 in Cohort 1: 1) Participants who were previously vaccinated with 2 or 3 doses of Sinopharm inactivated COVID-19 vaccine, with or without COVID-19 history; or 2) Participants who were previously vaccinated with 1 dose of Sinopharm inactivated COVID-19 vaccine and previously diagnosed with COVID-19. The interval between the date of last dose/COVID-19 diagnosis and the date of this study vaccination should be 3 to 24 months.

   For Cohort 2: 1) Participants who were previously vaccinated with 2 or 3 doses of mRNA COVID-19 vaccine (Comirnaty or mRNA-1273), with or without COVID-19 history; or 2) Participants who were previously vaccinated with 1 doses of mRNA COVID-19 vaccine (Comirnaty or mRNA-1273) and previously diagnosed with COVID-19; or 3) Participants who were previously not vaccinated with any COVID-19 vaccine and previously diagnosed with COVID-19. The interval between the date of last dose/COVID-19 diagnosis and the date of this study vaccination should be 3 to 24 months.
3. The participant and/or his legally acceptable representative can sign written ICF, and can fully understand the trial procedure, the risk of participating in the trial, and other interventions that can be selected if they do not participate in the trial;
4. The participant and/or his legally acceptable representative have the ability to read, understand, and fill in record cards;
5. Healthy participants or participants with pre-existing medical conditions who are in stable condition. The "pre-existing medical conditions" include but not limited to hypertension, diabetes, chronic cholecystitis and cholelithiasis, chronic gastritis that meet the described criteria. A stable medical condition is defined as disease not requiring significant change in therapy or no need for hospitalization as a consequence of worsening disease state for at least 3 months prior to enrollment;
6. Fertile men and women of childbearing potential voluntarily agree to take effective contraceptive measures from signing ICF to 6 months after the study vaccination; the pregnancy test results of women of childbearing potential are negative on screening.

Exclusion Criteria:

1. For Subgroup 1 in Cohort 1 only: Previously diagnosed with COVID-19.
2. Presence of fever within 3 days before the study vaccination;
3. A history of infection or disease related to severe acute respiratory syndrome (SARS), Middle East respiratory syndrome (MERS), or other disease corresponding use of immunosuppressants;
4. A history of allergic reactions to any vaccine or drug, such as allergy, urticaria, severe skin eczema, dyspnea, laryngeal edema, and angioneurotic edema;
5. A medical or family history of seizure, epilepsy, encephalopathy and psychosis;
6. Immunocompromised patients suffering from immunodeficiency diseases, important organ diseases, immune diseases (including Guillain-Barre Syndrome [GBS], systemic lupus erythematosus, rheumatoid arthritis, asplenia or splenectomy caused by any circumstances, and other immune diseases that may have an impact on immune response in the investigator's opinion), etc.;
7. Long-term use of immunosuppressant therapy or immunomodulatory drugs for ≥14 days within the first six months prior to enrollment. Whereas short-term (≤14 days) use of oral, inhaled and topical steroids are allowed;
8. Patients on antituberculosis therapy;
9. Presence of severe or uncontrollable cardiovascular diseases, or severe or uncontrollable disorders related to endocrine system, blood and lymphatic system, liver and kidney, respiratory system, metabolic and skeletal systems, or malignancies (skin basal cell carcinoma and carcinoma in-situ of cervix are exceptions and will not be excluded), such as severe heart failure, severe pulmonary heart disease, unstable angina, liver failure, or uremia;
10. Contraindications for intramuscular injection or intravenous blood sampling, including thrombocytopenia and other blood coagulation disorders;
11. Participants who received any immunoglobulin or blood products in the previous 3 months before enrollment, or plan to receive similar products during the study;
12. Participants who received other investigational drugs within 1 month before the study vaccination;
13. Participants who is at the acute state of disease, such as acute onset of chronic heart failure, acute sore throat, hypertensive encephalopathy, acute pneumonia, acute renal insufficiency, acute cholecystitis;
14. Participants received other drugs or vaccines used to prevent COVID-19, but participants previously received Sinopharm inactivated COVID-19 vaccine, Comirnaty or mRNA-1273 will not be excluded;
15. Participants vaccinated with influenza vaccine within 14 days or with other vaccines within 28 days before the study vaccination;
16. Those who donated blood or had blood loss (≥450 mL) within 3 months before the vaccination or plan to donate blood during the study period;
17. Those who are pregnant or breast-feeding or plan to be pregnant during the study period;
18. Those who plan to donate ovum or sperms during the study period;
19. Those who cannot follow the trial procedures, or cannot cooperate to complete the study due to planned relocation or long-term outing;
20. Those unsuitable for participating in the clinical trial as determined by the investigator because of other abnormalities that are likely to confuse the study results, or non-conformance with the maximal benefits of the participants;
21. Those who are tested positive for HIV in terms of serology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
GMT of nAb against Delta variant on Day 28 | Day 28 after the study vaccination
GMT of nAb against Omicron variant on Day 28 | Day 28 after the study vaccination

SECONDARY OUTCOMES:
GMT of nAb against Delta variant on Day 180 | Day 180 after the study vaccination
GMT of nAb against Omicron variant on Day 180 | Day 180 after the study vaccination
Number of IFN-γ positive (characterizing Th1) and IL-4 positive (characterizing Th2) T cell subsets on Day 28 | Day 28 after the study vaccination
Seroresponse rates of nAb to Delta variant on Day 28. | Day 28 after the study vaccination
  Seroresponse is defined as a change from below the low limit of quantitation [LLOQ] to equal to or above LLOQ, or a ≥4-fold rise if baseline is equal to or above LLOQ in nAb from Day0
Seroresponse rates of nAb to Omicron variant on Day 28. | Day 28 after the study vaccination
  Seroresponse is defined as a change from below the low limit of quantitation [LLOQ] to equal to or above LLOQ, or a ≥4-fold rise if baseline is equal to or above LLOQ in nAb from Day0
Incidence and severity of solicited AEs of SCTV01C from Day 0 to Day 7 | Day 0 to Day 7 after the study vaccination
Incidence and severity of all unsolicited AEs of SCTV01C from Day 0 to Day 28 | Day 0 to Day 28 after the study vaccination
Incidence and severity of SAEs and AESIs of SCTV01C within 180 days | Day 0 to Day 180 after the study vaccination
Incidence and severity of solicited AEs of SCTV01E from Day 0 to Day 7 | Day 0 to Day 7 after the study vaccination
Incidence and severity of all unsolicited AEs of SCTV01E from Day 0 to Day 28 | Day 0 to Day 28 after the study vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Al Kuwait Hospital (Al Baraha Hospital), Dubai, United Arab Emirates

REFERENCES:
- [Derived] Hannawi S, Yan L, Saifeldin L, Abuquta A, Alamadi A, Mahmoud SA, Hassan A, Zhang M, Gao C, Chen Y, Gai W, Xie L. Safety and immunogenicity of multivalent SARS-CoV-2 protein vaccines: a randomized phase 3 trial. EClinicalMedicine. 2023 Sep 8;64:102195. doi: 10.1016/j.eclinm.2023.102195. eCollection 2023 Oct. PMID 37731938
- [Derived] Wang R, Huang H, Yu C, Sun C, Ma J, Kong D, Lin Y, Zhao D, Zhou S, Lu J, Cao S, Zhang Y, Luo C, Li X, Wang Y, Xie L. A spike-trimer protein-based tetravalent COVID-19 vaccine elicits enhanced breadth of neutralization against SARS-CoV-2 Omicron subvariants and other variants. Sci China Life Sci. 2023 Aug;66(8):1818-1830. doi: 10.1007/s11427-022-2207-7. Epub 2022 Dec 30. PMID 36598621